CLINICAL TRIAL: NCT03333161
Title: Prematurity-Related Ventilatory Control (PRE-VENT): Role in Respiratory Outcomes Clinical Research Centers (CRC)
Brief Title: Prematurity Related Ventilatory Control (PRE-VENT) - Specific Aim 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Namasivayam Ambalavanan, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: UAB Neo 017; U01HL133536 (NIH)
Record Dates: First submitted 2017-11-02; First posted 2017-11-06 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Infant,Premature
Keywords: apnea of prematurity; bradycardia; hypoxemic episode; permissive hypercapnia
MeSH Terms: conditions — Premature Birth; Apnea; Bradycardia

STUDY DESIGN:
Intervention Model Description: The investigators will use the data from the 96 hours of intensive multiparametric physiologic monitoring at 2 weeks postnatal age. The first 24 hours of the data collection will be the baseline data, followed by evaluation of 3 interventions in a cross-over manner, with the initial intervention randomly assigned (computer-generated): Intervention 1 (24-48h of data), Intervention 2 (48-72h), and Intervention 3 (72-96h). The interventions will be to adjust transcutaneous carbondioxide measurements (TcCO2) up or down by 5 mm Hg, while maintaining TcCO2 within usual safe thresholds.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Higher TcCO2 (Experimental): The investigators will evaluate the effects of attempts to increase blood carbon dioxide levels within a narrow range of 5 mm Hg (well within the range of usual clinical practice) in a cross-over manner for 24 hours at a time, over a 4-day period, and use Cardiorespiratory Monitoring to evaluate control of breathing.
  The investigators will attempt to adjust PCO2 by 5 mm Hg higher from baseline (to max of 70 mm Hg), as long as pH is >7.2. The first 24 hours of the data collection will be the baseline data. Over the next 72 hours, the investigators will evaluate 3 interventions in a cross-over manner, with the initial intervention randomly assigned: Intervention 1 (24-48h of data; Increase TcCO2 by 5 mm Hg), Intervention 2 (48-72h; TcCO2 back to baseline), and Intervention 3 (72-96h; increase TcCO2 again by 5 mm Hg).
  Interventions: Diagnostic Test: Cardiorespiratory monitoring
- Lower TcCO2 (Active Comparator): The investigators will evaluate the effects of attempts to decrease blood carbon dioxide levels within a narrow range of 5 mm Hg (well within the range of usual clinical practice) in a cross-over manner for 24 hours at a time, over a 4-day period, and use Cardiorespiratory Monitoring to evaluate control of breathing.
  The investigators will attempt to adjust PCO2 by 5 mm Hg lower than baseline (to minimum of 40 mm Hg), as long as pH is <7.45.
  Interventions: Diagnostic Test: Cardiorespiratory monitoring

INTERVENTIONS:
Diagnostic Test: Cardiorespiratory monitoring — We will use high resolution physiologic monitoring of Heart Rate, Respiratory Rate, Pulse oximetry, (and near-infrared monitoring as well as microcapnography in selected infants) to evaluate control of breathing (apnea, bradycardia, desaturations).

SUMMARY:
To determine if late (at or beyond postnatal day 14) mild permissive hypercapnia is associated with reduction in apnea, bradycardia, and hypoxemic episodes and with improved stability of oxygenation.

DETAILED DESCRIPTION:
Preterm infants who remain intubated or on nasal mechanical ventilation (IMV) at 14 days postnatal age, meet blood gas criteria, have transcutaneous carbondioxide (TcCO2) monitoring with TcCO2 values that trend and correlate appropriately with PaCO2, and are not judged too unstable by Attending neonatologist will qualify.

The investigators will use the data from the 96 hours of intensive multiparametric physiologic monitoring at 2 weeks postnatal age.

The first 24 hours of data collection will be the baseline data. Over the next 72 hours, the investigators will evaluate 3 interventions in a cross-over manner with the initial intervention randomly assigned: Intervention 1 (24-48h of data), Intervention 2 (48-72h of data) and Intervention 3 (72-96h of data).

ELIGIBILITY:
Inclusion Criteria:

1. Inborn infants weighing 401-1,000 grams on admission and/or 22w 0/7d to 28w 6/7d (<29 weeks) inclusive completed weeks of gestation
2. Infants eligible for full care and resuscitation as necessary, and surviving beyond 24 h of age
3. Enrollment in main study protocol (Aim 1 of PreVENT Apnea) at <1 week post-natal age
4. Informed consent from parent/guardian
5. This study will enroll the subset of infants from Aim 1 who are still intubated or on nasal IMV at 2 weeks postnatal age, meet blood gas criteria (arterial or capillary arterialized blood gas values done q12-24h, as most infants do not have an arterial line at 2 weeks: pH >7.25, PaCO2 >40 mm Hg), have TcCO2 monitoring with TcCO2 values that trend and correlate appropriately with PaCO2, and are not judged too unstable by the Attending neonatologist.

Exclusion Criteria:

1. Refusal or withdrawal of consent
2. Major congenital malformations (e.g., not including patent ductus arteriosus, small hernia)

Ages: 1 Day to 15 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Hypoxemic episode | During 24 hour time periods with targeted transcutaneous carbondioxide (TcCO2)
  Hypoxemic episode defined as as oxygen saturation by pulse oximetry (SpO2 )<85% for >10 seconds

SECONDARY OUTCOMES:
Bradycardic episode | During 24 hour time periods with targeted TcCO2
  Bradycardic episode defined as heart rate (HR) <100/min for >10 seconds
Apnea episodes | During 24 hour time periods with targeted TcCO2
  Apnea defined as Respiratory Rate (RR)=0 for >20 seconds, or RR=0 for >10 seconds + SpO2 <85% or HR <100/min
Hypoxemic time | During 24 hour time periods with targeted TcCO2
  Hypoxemic time defined as duration of time with SpO2 <85%
Bronchopulmonary dysplasia (BPD) | 36 weeks PMA
  BPD defined using physiologic definition at 36w Post-Menstrual Age (PMA)

CONTACTS AND LOCATIONS:
Overall Officials: Namasivayam Ambalavanan, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- Regional Neonatal ICU and CCN, University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Travers CP, Carlo WA, Nakhmani A, Laney D, Chahine RA, Aban I, Ambalavanan N. Late permissive hypercapnia and respiratory stability among very preterm infants: a pilot randomised trial. Arch Dis Child Fetal Neonatal Ed. 2023 Sep;108(5):530-534. doi: 10.1136/archdischild-2022-325166. Epub 2023 Mar 13. PMID 36914233

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-26): https://cdn.clinicaltrials.gov/large-docs/61/NCT03333161/Prot_SAP_000.pdf